CLINICAL TRIAL: NCT03574948
Title: Multicentric, Double-blind, Placebo Controlled Clinical Trial With 5-hydroxytryptophan (5-HTP) in Patients With Inflammatory Bowel Disease in Clinical and Biologic Remission: Effect on Fatigue Scores
Brief Title: 5-HTP in Patients With IBD in Clinical and Biologic Remission:Effect on Fatigue Scores
Acronym: TRP-IBD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-005059-10
Record Dates: First submitted 2018-06-22; First posted 2018-07-02 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-01

CONDITIONS: Crohn Disease; Ulcerative Colitis; Fatigue; Remission
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Fatigue | interventions — 5-Hydroxytryptophan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-HTP (Experimental): 8 weeks active substance 5-HTP (2 x 100 mg per day)
  Interventions: Drug: 5-HTP
- placebo oral capsule (Placebo Comparator): 8 weeks placebo (2 x 1 capsule per day)
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: 5-HTP — 8 weeks active substance 5-HTP (2 x 100mg per day)
  Other Names: Levotonine
  Arms: 5-HTP
Drug: Placebo oral capsule — 8 weeks placebo (2 x 1 caps per day)
  Other Names: placebo
  Arms: placebo oral capsule

SUMMARY:
This placebo cross-over trial aims to study the effect of the oral intake of an essential amino-acid 5-OH tryptophan, the precursor of serotonin, on the fatigue scores in IBD patients in deep clinical and biological remission.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female and aged 18 to 60 yrs (inclusive)
* The subject has a documented Crohn's disease or ulcerative colitis
* The subject is, in the opinion of the investigator, capable of understanding and complying protocol requirements
* The subject is in clinical remission over last 3 months (based on physician global assessment)
* The subject is in clinical remission at day 0 based on validated scores (SCCAI ≤ 2 for ulcerative colitis or Harvey Bradshaw index ≤ 4 for Crohn's disease).
* The subject reports fatigue on a quantified scale (visual analogue scale 0 - 10) of 5 or more
* The subject is treated with biologicals and/or immunosuppressives since at least 6 months with stable dose over last 3 months
* The subject is in biologic remission at day 0: CRP < 10 mg/l and faecal calprotectin value < 250 mg/kg

Exclusion Criteria:

* The subject has a clinical validated depression
* The subject is taking antidepressives or neuroleptics
* The subject has a psychiatric comorbidity
* The subject has important comorbidities: cardiovascular disease, obstructive lung pathology, neoplasia or other
* The subject has a documented Anemia (based on lab results including Hb < 12-13 g/dl respectively for saturation index < 20%, Vit B12 < 148 pmol/L or folic acid < 6 nmol/L)
* The subject has a documented hypothyreoidea (documented by a recent lab result including TSH)
* The subject reports an infection within 2 weeks before inclusion
* The subject reports any change in IBD medication (biologicals and immunosuppressives) in the last 12 weeks before inclusion
* The subject was treated with oral corticosteroids during the last 8 weeks before enrolment
* The subject reports an ongoing pregnancy or breastfeeding
* The subject has a history of lymphoproliferative disease or cancer other than basocellular skin cancer
* The subject underwent surgery in the past 12 weeks prior to the screening visit
* The subject reports a history of clinically significant drug abuse (defined as any illicit drug use) or alcohol abuse within 1 year prior to inclusion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) after intervention | weekly, 16 weeks
  Patients are asked to indicate their fatigue level on a VAS-scale from 0 to 10, where 0 represents no fatigue and where 10 indicates the patient suffers from severe fatigue.

SECONDARY OUTCOMES:
Changes in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) score | week 0, week 8 and week 16
  The questionnaire is a self-assessment that need to be completed without external help. The FACIT-F questionnaire measures the fatigue of the patient and will be filled in at week 0, week 8 and week 16. The FACIT Fatigue scale ranges from 0 to 52, with high scores indicating higher levels of fatigue.
Changes in short Depression Anxiety and Stress Scale (DASS21) | week 0, week 8 and week 16
  The questionnaire is a self-assessment that need to be completed without external help. The DASS questionnaire measures depression and anxiety and will be filled in at week 0, week 8 and week 16. The questionnaire contains 7 items per scale, the maximum score for depression, anxiety and stress will be 21. The higher the score of the questionnaire, the more the patient suffers from depression, anxiety and stress.
Change in Adapted International Physical Activity Questionnaire (IPAQ) | week 0, week 8 and week 16
  The adapted IPAQ questionnaire measures the physical activity and will be filled in at week 0, week 8 and week 16.
Changes in serum 5-HydroxyTryptophane (5-HTP) by treatment | Week 0, week 8 and week 16
  The possible effect of Levotonine administration on the serum 5-HTP levels will be measured.
Changes in serum 5-hydroxyindoleacetic acid by treatment | Week 0, week 8 and week 16
  The possible effect of Levotonine administration on the serum 5-hydroxyindoleacetic levels will be measured.
Changes in serum serotonin levels by treatment | Week 0, week 8 and week 16
  The possible effect of Levotonine administration on the serum serotonin levels will be measured.
Changes in serum melatonin levels by treatment | Week 0, week 8 and week 16
  The possible effect of Levotonine administration on the serum melatonin levels will be measured.
Changes in faecal microbiome/metabolome | Week 0, week 8 and week 16
  since the intestinal bacteria can process tryptophane, changes in the faecal microbiome/metabolome can be possibly caused by the administration of levotonine.

CONTACTS AND LOCATIONS:
Overall Officials: Martine De Vos, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (13):
- Belgium (13):
  - AZ Imelda, Bonheiden
  - CHU Saint-Pièrre, Brussels
  - UCL Saint-Luc, Brussels
  - ULB Erasme, Brussels
  - UZ Brussel, Brussels
  - Ghent University Hospital, Ghent
  - AZ Maria Middelares, Ghent
  - AZ Sint-Lucas, Ghent
  - UZ Leuven, Leuven
  - CHU Liège, Liège
  - CHU Namur, Namur
  - AZ Damiaan, Ostend
  - AZ Nikolaas, Sint-Niklaas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Truyens M, Lobaton T, Ferrante M, Bossuyt P, Vermeire S, Pouillon L, Dewint P, Cremer A, Peeters H, Lambrecht G, Louis E, Rahier JF, Dewit O, Muls V, Holvoet T, Vandermeulen L, Peeters A, Gonzales GB, Bos S, Laukens D, De Vos M. Effect of 5-Hydroxytryptophan on Fatigue in Quiescent Inflammatory Bowel Disease: A Randomized Controlled Trial. Gastroenterology. 2022 Nov;163(5):1294-1305.e3. doi: 10.1053/j.gastro.2022.07.052. Epub 2022 Aug 6. PMID 35940251